CLINICAL TRIAL: NCT05894551
Title: Investigation of the Changing of Quadriceps Angle in Static and Dynamic Postures in Healthy Adults and Its Relation With Physical Parameters
Brief Title: Q Angle in Static and Dynamic Postures
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Asssistant professor, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC_dynamicqangle
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Quadriceps Muscle; Orthopedic Disorder
Keywords: q angle; dynamic q angle; lower extremity function
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy participants: Volunteers aged 18-25 years, healthy individuals without any spinal or neurologic injury and any injury leading to ligament, muscle or bone defect in their lower extremities
  Interventions: Other: Evaluation of q angles different positions; Other: Physical examination; Other: Functional mobility assessment

INTERVENTIONS:
Other: Evaluation of q angles different positions — Q angle evaluation in two different static postures (upright and supine position) and dynamic posture during the midstance phase of the gait
Other: Physical examination — With goniometric evaluations, the femoral anteversion angle will be measured. Pelvis width and thigh length will be measured with a tape measure. Quadriceps muscle strength, hamstring muscle strength, Hip abduction, adduction, internal and external rotation and extension muscle strength will be measured with hand-held dynamometer.
  Joint mobility will be assessed with the Beighton score and foot posture will be evaluated with the foot posture index-6 (FPI-6).
Other: Functional mobility assessment — 10-meter walking test will be conducted to understand functional mobility.

SUMMARY:
The Q angle, also known as the quadriceps angle, is defined as the angle formed between the quadriceps muscles and the patella tendon. It was first described by Brattstrom in 1964 (1). The Q angle is the angle between the line extending from the anterior superior of the spina iliaca to the midpoint of the patella and the line extending from the midpoint of the patella to the tuberositas tibia (2). Normally, this angle is between 8-14 degrees in men and 11-20 degrees in women. Any alignment change that increases the Q angle is thought to increase the lateral force on the patella.

The Q angle is generally evaluated in static postures in the literature. The Q angle value varies according to the patient's gender, the contractility of the quadriceps, and the patient's posture (standing or supine) (3).

Q angle was evaluated in a static posture with a standard goniometer or computerized biophotogrammetry (4) Q angle changes with the forces applied by dynamic structures. It is insufficient to evaluate only in a static posture. Therefore, the aim of this study is to examine the effect of dynamic structures on the Q angle using 2D gait analysis (video) and to detect the early signs of deviation of changes in the q angle.

DETAILED DESCRIPTION:
The Q angle is a very important tool in evaluating the function of the knee joint and describing the biomechanical alignment and function of the lower extremity (5). Abnormal values may cause joint problems later on, and in some cases, may affect the quadriceps reflex time, causing subluxation of the patella or an increased risk of developing anterior cruciate ligament ACL injury (5). For this reason, the Q angle is routinely and regularly used as an evaluation parameter when diagnosing many knee-related problems, including anterior knee pain, osteoarthritis, and degenerative knee disorders. When evaluated correctly, it provides very useful information about the alignment of the pelvis, legs and feet (6-8).

Therefore, determining the Q angle is very important, especially for athletic and physically active patients (9). In most studies, the Q angle was measured using a goniometer or with a modified goniometer (10-12). Biedert et al. by radiography (3). Braz et al. determined the Q angle with digital photogrammetry (13). In the literature, the q angle was generally evaluated in the supine or standing position (14). Higher Q angle values have been reported when transitioning from the supine position to the standing position (15). The increased Q angle while standing has been attributed to changes in lower extremity alignment due to weight bearing. In studies in the literature, the q angle was generally evaluated in static postures. In an ideal postural alignment, there should be a dynamic balance between muscles, joints and skeletal structures (16-17). Not only static structures but also dynamic structures are responsible for problems related to the alignment of the patella. For this reason, it is important to know the changes in the q angle not only in static postures but also in dynamic postures. Evaluation in correct postures is essential for diagnosis, planning and follow-up of the development and results of physical therapy (16).

The primary aim of this study was to report the prevalence and normative reference values of the q angle in the midstance phase of gait using 2D analysis (video).

The secondary aim of this study is to examine the variation of q angles during the midstance phase gait with Q angle values in static postures.

The tertiary aim of this study is to examine the relationship of q angles with different parameters such as age, gender, BMI, lower extremity strength, and hypermobility.

Demographic information (age, weight, height, etc.) will be obtained from healthy volunteers included in the study. As primary outcome measures, q-angles will be measured in static posture (supine and standing) and dynamic posture (with video analysis). Markers will be placed on the relevant places (SIAS, Patella middle and tuberositas tibia). Afterward, the video recordings will be played in slow motion and the evaluators will pause the video during the mid-stance phases of the gait, and the q-angles will be determined with the two-dimensional video analysis software (Kinoveav.0.8.15).

As secondary outcome measures, pelvis width and thigh length with a tape measure and femoral anteversion goniometer with quadriceps muscle strength, hamstring muscle strength, Hip abduction, adduction, internal and external rotation and extension muscle strength with hand-held dynamometer, joint mobility with Beighton score, foot posture index and functionality will be evaluated by walking 8 meters.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-25
* being volunteer
* not have any condition that may affect cooperation

Exclusion Criteria:

* Individuals with any injury to their lower extremities that cause ligament, muscle or bone defect and any spinal or neurological injury
* individuals diagnosed with any knee disorder such as fracture, acute or chronic knee pain, patella dislocation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers aged 18-25 years, healthy individuals without any spinal or neurologic injury and any injury leading to ligament, muscle or bone defect in their lower extremities.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Q angle | baseline
  Q angle measurement in three different position; in supine, standing and midstance phase during gait. The static and dynamic positions of the participants will be recorded as a photo and frame from video recording, then the measurements will be conducted with 2-dimensions movement analysis software. The unit of measurement will be recorded in angle degree.

SECONDARY OUTCOMES:
Pelvic width | baseline
  Pelvic width will be measured with a tape and the unit of measurement will be recorded in centimeters.
Thigh length | baseline
  It will be measured with a tape and the unit of measurement will be recorded in centimeters.
Femoral anteversion angle | baseline
  The femoral anteversion angle will be measured with goniometer. The normal angle is +10 degrees, with a range of -3 to +20 degrees. The unit of measurement will be recorded in angle degree.
Lower extremity muscle strength | baseline
  Quadriceps muscle strength, hamstring muscle strength, Hip abduction, adduction, internal and external rotation and extension muscle strength will be measured with hand-held dynamometer. The unit of measurement will be recorded in libre.
Beighton score | baseline
  Joint mobility will be assessed with the Beighton score. Simple actions like bending your pinky (little) finger backward to evaluate the joint angle are involved. A nine-point scoring system is used for the Beighton score. The joints are more flexible the higher your score.
Foot posture index-6 | baseline
  Foot posture will be evaluated with the foot posture index-6 (FPI-6). The FPI-6 is a rapid, accurate diagnostic tool that rates foot posture using predetermined criteria and an easy scale. It is used to determine how pronated, neutral, or supinated a foot is. Pronated postures are given a positive value, the higher the value the more pronated.
  Supinated features are given a negative value, the more negative the value the more supinated.
  For a neutral foot the final FPI aggregate score should lie somewhere around zero.
10-meter walking test | baseline
  10-meter walking test will be conducted to understand functional mobility. The 10 Metre Walk Test is a performance indicator used to evaluate walking speed over a brief distance in meters per second. To assess functional mobility, gait, and vestibular function, it can be used. The cut-off values like that; Household Ambulator <0.40 m/s; Limited Community Ambulator 0.40 to <0.80 m/s; Community Ambulator ≥0.80 m/s. the unit of measurement will be recorded in second.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa, Istanbul, Istanbul
  - Hatay Mustafa Kemal University, Hatay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BRATTSTROEM H. SHAPE OF THE INTERCONDYLAR GROOVE NORMALLY AND IN RECURRENT DISLOCATION OF PATELLA. A CLINICAL AND X-RAY-ANATOMICAL INVESTIGATION. Acta Orthop Scand Suppl. 1964;68:SUPPL 68:1-148. No abstract available. PMID 14171734
- [Background] Merchant AC, Fraiser R, Dragoo J, Fredericson M. A reliable Q angle measurement using a standardized protocol. Knee. 2020 Jun;27(3):934-939. doi: 10.1016/j.knee.2020.03.001. Epub 2020 Apr 12. PMID 32295725
- [Background] Biedert RM, Warnke K. Correlation between the Q angle and the patella position: a clinical and axial computed tomography evaluation. Arch Orthop Trauma Surg. 2001 Jun;121(6):346-9. doi: 10.1007/s004020000239. PMID 11482469
- [Background] Iunes DH, Castro FA, Salgado HS, Moura IC, Oliveira AS, Bevilaqua-Grossi D. Confiabilidade intra e interexaminadores e repetibilidade da avaliação postural pela fotogrametria. Rev Bras Fisioter. 2005;9(3):327-334.
- [Background] Khasawneh RR, Allouh MZ, Abu-El-Rub E. Measurement of the quadriceps (Q) angle with respect to various body parameters in young Arab population. PLoS One. 2019 Jun 13;14(6):e0218387. doi: 10.1371/journal.pone.0218387. eCollection 2019. PMID 31194851
- [Background] Daneshmandi H, Saki F, Shahheidari S, Khoori A. Lower extremity Malalignment and its linear relation with Q angle in female athletes. 3rd World Conf Educ Sci-2011. 2011;15: 3349-3354.
- [Background] Nguyen AD, Boling MC, Levine B, Shultz SJ. Relationships between lower extremity alignment and the quadriceps angle. Clin J Sport Med. 2009 May;19(3):201-6. doi: 10.1097/JSM.0b013e3181a38fb1. PMID 19423972
- [Background] Almeida GP, Silva AP, Franca FJ, Magalhaes MO, Burke TN, Marques AP. Q-angle in patellofemoral pain: relationship with dynamic knee valgus, hip abductor torque, pain and function. Rev Bras Ortop. 2016 Feb 9;51(2):181-6. doi: 10.1016/j.rboe.2016.01.010. eCollection 2016 Mar-Apr. PMID 27069887
- [Background] Yilmaz A, Kabadayi M, Mayda M, Çavusoglu G, Tasmektepligi M. Analysis of Q Angle Values of Female Athletes from Different Branches. Sci Mov Heal. 2017;17: 141-146.
- [Background] Omololu BB, Ogunlade OS, Gopaldasani VK. Normal Q-angle in an adult Nigerian population. Clin Orthop Relat Res. 2009 Aug;467(8):2073-6. doi: 10.1007/s11999-008-0637-1. Epub 2008 Nov 26. PMID 19034592
- [Background] Greene CC, Edwards TB, Wade MR, Carson EW. Reliability of the quadriceps angle measurement. Am J Knee Surg. 2001 Spring;14(2):97-103. PMID 11401177
- [Background] Raveendranath R, Nachiket S, Sujatha N, Priya R, Rema D. Bilateral Variability of the Quadriceps Angle (Q angle) in an Adult Indian Population. Iran J Basic Med Sci. 2011 Sep;14(5):465-71. PMID 23493777
- [Background] Braz RG, Carvalho GA. Relationship between quadriceps angle (Q) and plantar pressure distribution in football players. Rev Bras Fisioter. 2010 Jul-Aug;14(4):296-302. Epub 2010 Sep 3. English, Portuguese. PMID 20949230
- [Background] Choudhary R, Malik M, Aslam A, Khurana D, Chauhan S. Effect of various parameters on Quadriceps angle in adult Indian population. J Clin Orthop Trauma. 2019 Jan-Feb;10(1):149-154. doi: 10.1016/j.jcot.2017.11.011. Epub 2017 Nov 23. PMID 30705551
- [Background] Guerra JP, Arnold MJ, Gajdosik RL. Q angle: effects of isometric quadriceps contraction and body position. J Orthop Sports Phys Ther. 1994 Apr;19(4):200-4. doi: 10.2519/jospt.1994.19.4.200. PMID 8173567
- [Background] Rosario L.R. What is posture? a review of the literature in search of a definition. EC Orthopaedics. 2017;6(3):111-133.
- [Background] Sacco I.C.N., AlIbert S., Queiroz B.W., Pripas D., KlelIng I., Kimura A.A. Reliability of photogrammetry in relation to goniometry for postural lower limb assessment. Rev Bras Fisioterpp. 2007;11(5):411-417.